CLINICAL TRIAL: NCT04683744
Title: Facilitators and Barriers to Cancer Screening: Stakeholder Perspectives on Implementation
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Principal Investigator, Indiana University
Other Study IDs: 2012926551; CDR-2018C3-14715 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Screening
Keywords: decision aid; decision making; COVID-19; risk communication; colorectal neoplasm; electronic health records
MeSH Terms: conditions — COVID-19; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare system leadership, providers, and staff: Leadership, providers, and staff at the study team's affiliated health systems.
  Interventions: Other: Semi-structured interviews-Health system
- Patients receiving primary care at the study team's affiliated health systems: Patients who had a least one primary care visit during the past 24 months at the study team's affiliated health care systems.
  Interventions: Other: Semi-structured interviews-Patients

INTERVENTIONS:
Other: Semi-structured interviews-Patients — The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
  Groups: Patients receiving primary care at the study team's affiliated health systems
Other: Semi-structured interviews-Health system — The interview guide will consist of questions to elicit thoughts from health system leadership, providers, and staff about implementing decision aids, provider notifications, and cancer risk assessments in their health center or healthcare system. The questions may be specific to colorectal cancer screening or more generally about other cancer screenings. The investigators may also ask questions about cancer screening initiatives their health center or healthcare system engaged in during the COVID-19 pandemic.
  Groups: Healthcare system leadership, providers, and staff

SUMMARY:
The rate of screening for colorectal cancer (CRC) in the U.S. remains low (under 65%), meaning that thousands of people die of colorectal cancer unnecessarily. Colorectal cancer screening tests range from more invasive and very sensitive for polyps and cancer (colonoscopy) to less invasive and less sensitive (e.g., fecal immunochemical testing (FIT)). Screening rates go up when patients consider all these tests, not just colonoscopy. Informing patients about their options for CRC screening could produce higher quality decisions, improve the match between patient preferences and tests performed, and increase uptake of CRC screening. Decision aids (DAs) are a promising tool for accomplishing this goal. Also, precision CRC prevention - providing information about an individual's specific risk for CRC - has great promise to increase uptake and improve decision making.

Unfortunately, the COVID-19 pandemic is causing severe challenges to providing CRC screening and other prevention services. Health systems are trying to adapt, but these efforts have only begun and are poorly understood. Moreover, patient perceptions of disease risk and risk from COVID-19 are unknown.

DETAILED DESCRIPTION:
The study team will engage with the leadership, staff, and providers in the study team's partner healthcare systems, to identify facilitators and barriers to implementing patient decision aids and provider notifications as well as cancer risk assessment tools, for colorectal cancer screening, and for other evidence-based cancer screening during the COVID pandemic and, potentially, after the conclusion of the pandemic.

At the conclusion of the study, the investigators will have extensive information regarding how best to provide decision aids through an electronic health record (EHR) portal, with or without personalized information, and to deliver provider notifications, which can guide broader implementation.

The study will involve interviews with staff and providers at the study team's partner healthcare systems to identify facilitators and barriers to implementing decision aids and provider notifications for colorectal cancer screening.

Also, the investigators will interview patients to identify perceptions of prevention during the COVID-19 pandemic including risk perception and barriers to screening, perceptions of risk from both the pandemic and disease, and patient cancer screening and risk prevention behaviors engaged in or postponed during the pandemic and patient rationales for their decisions. This part of the study will suggest potentially promising approaches for providing prevention and disease management during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

Health system participants will be eligible if:

* they are employed by one of the study team's partner healthcare systems.

Patient participants will be eligible if:

* they have had a primary care visit during the past 24 months
* they have completed cancer screening during the past 5 years prior to 2020 for breast, cervical or lung cancer as noted in the electronic health record (EHR)
* age 50 years or older
* speaks English
* accessible by phone.

Exclusion Criteria:

Patients will be excluded if:

* they did not complete any cancer screening for breast, colon, cervical, or lung cancer during the past 5 years prior to 2020
* did not complete a primary care visit at a partner healthcare system during the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be health system primary care patients, and health system leadership, providers, or staff involved in primary care.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schwartz, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufman HW, Chen Z, Niles J, Fesko Y. Changes in the Number of US Patients With Newly Identified Cancer Before and During the Coronavirus Disease 2019 (COVID-19) Pandemic. JAMA Netw Open. 2020 Aug 3;3(8):e2017267. doi: 10.1001/jamanetworkopen.2020.17267. PMID 32749465
- [Background] Castanon A, Rebolj M, Pesola F, Sasieni P. Recovery strategies following COVID-19 disruption to cervical cancer screening and their impact on excess diagnoses. Br J Cancer. 2021 Apr;124(8):1361-1365. doi: 10.1038/s41416-021-01275-3. Epub 2021 Feb 9. PMID 33558708
- [Background] Chen RC, Haynes K, Du S, Barron J, Katz AJ. Association of Cancer Screening Deficit in the United States With the COVID-19 Pandemic. JAMA Oncol. 2021 Jun 1;7(6):878-884. doi: 10.1001/jamaoncol.2021.0884. PMID 33914015
- [Background] Alkatout I, Biebl M, Momenimovahed Z, Giovannucci E, Hadavandsiri F, Salehiniya H, Allahqoli L. Has COVID-19 Affected Cancer Screening Programs? A Systematic Review. Front Oncol. 2021 May 17;11:675038. doi: 10.3389/fonc.2021.675038. eCollection 2021. PMID 34079764
- [Background] Czeisler ME, Marynak K, Clarke KEN, Salah Z, Shakya I, Thierry JM, Ali N, McMillan H, Wiley JF, Weaver MD, Czeisler CA, Rajaratnam SMW, Howard ME. Delay or Avoidance of Medical Care Because of COVID-19-Related Concerns - United States, June 2020. MMWR Morb Mortal Wkly Rep. 2020 Sep 11;69(36):1250-1257. doi: 10.15585/mmwr.mm6936a4. PMID 32915166
- [Background] Findling MG, Blendon RJ, Benson JM. Delayed Care with Harmful Health Consequences-Reported Experiences from National Surveys During Coronavirus Disease 2019. JAMA Health Forum. 2020 Dec 1;1(12):e201463. doi: 10.1001/jamahealthforum.2020.1463. No abstract available. PMID 36218479
- [Background] Park S, Stimpson JP. Trends in Self-reported Forgone Medical Care Among Medicare Beneficiaries During the COVID-19 Pandemic. JAMA Health Forum. 2021 Dec 30;2(12):e214299. doi: 10.1001/jamahealthforum.2021.4299. eCollection 2021 Dec. PMID 35977302
- [Background] Lieneck C, Herzog B, Krips R. Analysis of Facilitators and Barriers to the Delivery of Routine Care during the COVID-19 Global Pandemic: A Systematic Review. Healthcare (Basel). 2021 May 1;9(5):528. doi: 10.3390/healthcare9050528. PMID 34062813
- [Background] Aitken M, Kleinrock M. Shifts in Healthcare Demand, Delivery and Care During the COVID-19 Era. Published online 2020. https://www.iqvia.com/insights/the-iqvia-institute/covid-19/shifts-in-healthcare-demand-delivery-and-care-during-the-covid-19-era
- [Background] Powell RE, Henstenburg JM, Cooper G, Hollander JE, Rising KL. Patient Perceptions of Telehealth Primary Care Video Visits. Ann Fam Med. 2017 May;15(3):225-229. doi: 10.1370/afm.2095. PMID 28483887
- [Background] Price ST, Mainous AG, Rooks BJ. Survey of cancer screening practices and telehealth services among primary care physicians during the COVID-19 pandemic. Prev Med Rep. 2022 Mar 17;27:101769. doi: 10.1016/j.pmedr.2022.101769. eCollection 2022 Jun. PMID 35313453
- [Background] Basu P, Alhomoud S, Taghavi K, Carvalho AL, Lucas E, Baussano I. Cancer Screening in the Coronavirus Pandemic Era: Adjusting to a New Situation. JCO Glob Oncol. 2021 Mar;7:416-424. doi: 10.1200/GO.21.00033. PMID 33784177
- [Background] Cancino RS, Su Z, Mesa R, Tomlinson GE, Wang J. The Impact of COVID-19 on Cancer Screening: Challenges and Opportunities. JMIR Cancer. 2020 Oct 29;6(2):e21697. doi: 10.2196/21697. PMID 33027039
- [Background] Horn DM, Haas JS. Expanded Lung and Colorectal Cancer Screening - Ensuring Equity and Safety under New Guidelines. N Engl J Med. 2022 Jan 13;386(2):100-102. doi: 10.1056/NEJMp2113332. Epub 2022 Jan 8. No abstract available. PMID 34995027
- [Background] Gorin SNS, Jimbo M, Heizelman R, Harmes KM, Harper DM. The future of cancer screening after COVID-19 may be at home. Cancer. 2021 Feb 15;127(4):498-503. doi: 10.1002/cncr.33274. Epub 2020 Nov 10. PMID 33170520
- [Background] Frey B. Snowball Sampling. In: The SAGE Encyclopedia of Educational Research, Measurement, and Evaluation. 2018. https://dx.doi.org/10.4135/9781506326139.n636
- [Background] Beebe J. Rapid Qualitative Inquiry: A Guide to Team Based Assessment.; 2014.
- [Background] Gale RC, Wu J, Erhardt T, Bounthavong M, Reardon CM, Damschroder LJ, Midboe AM. Comparison of rapid vs in-depth qualitative analytic methods from a process evaluation of academic detailing in the Veterans Health Administration. Implement Sci. 2019 Feb 1;14(1):11. doi: 10.1186/s13012-019-0853-y. PMID 30709368
- [Background] Nevedal AL, Reardon CM, Opra Widerquist MA, Jackson GL, Cutrona SL, White BS, Damschroder LJ. Rapid versus traditional qualitative analysis using the Consolidated Framework for Implementation Research (CFIR). Implement Sci. 2021 Jul 2;16(1):67. doi: 10.1186/s13012-021-01111-5. PMID 34215286
- [Background] Taylor B, Henshall C, Kenyon S, Litchfield I, Greenfield S. Can rapid approaches to qualitative analysis deliver timely, valid findings to clinical leaders? A mixed methods study comparing rapid and thematic analysis. BMJ Open. 2018 Oct 8;8(10):e019993. doi: 10.1136/bmjopen-2017-019993. PMID 30297341
- See also: Epic Health Research Network. Preventive Cancer Screenings during COVID-19 Pandemic. — https://www.ehrn.org/wp-content/uploads/Preventive-Cancer-Screenings-during-COVID-19-Pandemic.pdf
- See also: Centers for Medicare and Medicaid Centers for Medicare and Medicaid Services (CMS). Medicare telemedicine snapshot: Medicare claims and encounter data: March 1, 2020 to February 28, 2021. Received by September 9, 2021. — https://www.cms.gov/files/document/medicare-telemedicine-snapshot.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthcare system: we used snowball sampling to identify leadership, providers, and clinical staff involved in cancer screening, primary care and prevention. We interviewed 20 key informants in January-July 2021 and re-interviewed 11 of them in January-March 2022.
  Patients: we interviewed patients (screened and not screened) who were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020. Interviews were conducted from August 2021 through February 2022.
Pre-assignment Details: One patient that was consented, enrolled, and interviewed was removed from the study after review of data by PI and key research members concluded that the patient had undergone a diagnostic rather than screening procedure.
Groups:
- Not Screened Patients: Patients who had a least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020, and did NOT complete the screening they were selected for at time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
- Screened Patients: Patients who had at least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020 and did completed the screening they were selected for at time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
Period: Overall Study
Arm/Group | Healthcare System Leadership, Providers, and Staff | Not Screened Patients | Screened Patients
Started (Health system: approached for interview via email Patients: recruitment letter mailed) | 20 (Health System Participants Approached: 27; Unable to contact: 6; Declined to participate: 1) | 29 (Letters mailed: 227; Assessed eligibility: 86; Not eligible: 44; Declined to participate: 13) | 33 (Letters mailed: 106; Assessed eligibility: 47; Not eligible: 10; Declined to participate: 4)
Interview #1 | 20 | 29 | 33
Interview #2 | 11 | 0 (Patients completed one interview only) | 0 (Patients completed one interview only)
Completed | 20 | 29 | 32
Not Completed | 0 | 0 | 1
Not completed — withdrawn (determined not eligible after enrollment) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Not Screened Patients: Patients who were due for cancer screening (breast, cervical, colorectal or lung cancer) between April-July 2020, however had not completed the screening they were selected for at time of interview.
- Screened Patients: Patients who were due for cancer screening (breast, cervical, colorectal or lung cancer) between April-July 2020 and had completed the screening they were selected for at time of interview.
- Health System Participants: Leadership, providers, and clinical staff involved in cancer screening, primary care, and prevention at two affiliated health systems.
- Total: Total of all reporting groups
Arm/Group | Not Screened Patients | Screened Patients | Health System Participants | Total
Number analyzed (Participants) | 29 | 32 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic-age data for health system participants was not collected at baseline.
  years
    number analyzed (Participants) | 29 | 32 | 0 | 61
    (all) | 56.1 (15.1) | 56.2 (14.5) |  | 56.1 (14.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Demographic-sex/gender data for health system participants was not collected at baseline.
  Participants
    Female: number analyzed (Participants) | 29 | 32 | 0 | 61
    Female | 24 | 23 |  | 47
    Male: number analyzed (Participants) | 29 | 32 | 0 | 61
    Male | 4 | 9 |  | 13
    Other: number analyzed (Participants) | 29 | 32 | 0 | 61
    Other | 1 | 0 |  | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographic-race and ethnicity data for Health system participants was not collected at baseline.
  Participants
    White: number analyzed (Participants) | 29 | 32 | 0 | 61
    White | 17 | 16 |  | 33
    Black or African American: number analyzed (Participants) | 29 | 32 | 0 | 61
    Black or African American | 11 | 13 |  | 24
    Other: number analyzed (Participants) | 29 | 32 | 0 | 61
    Other | 1 | 3 |  | 4
    Hispanic/Latino: number analyzed (Participants) | 29 | 32 | 0 | 61
    Hispanic/Latino | 0 | 0 |  | 0
Living Situation [Count of Participants; unit: Participants] — Population: Living situation data will not be collected for health system participants.
  Participants
    Never Married: number analyzed (Participants) | 29 | 32 | 0 | 61
    Never Married | 7 | 9 |  | 16
    Married/Living with a Partner: number analyzed (Participants) | 29 | 32 | 0 | 61
    Married/Living with a Partner | 14 | 13 |  | 27
    Divorced: number analyzed (Participants) | 29 | 32 | 0 | 61
    Divorced | 3 | 4 |  | 7
    Separated: number analyzed (Participants) | 29 | 32 | 0 | 61
    Separated | 0 | 1 |  | 1
    Widowed: number analyzed (Participants) | 29 | 32 | 0 | 61
    Widowed | 5 | 5 |  | 10
Highest Level of Education [Count of Participants; unit: Participants] — Population: Education level will not be collected for health system participants.
  Participants
    Less than high school diploma: number analyzed (Participants) | 29 | 32 | 0 | 61
    Less than high school diploma | 2 | 3 |  | 5
    High school graduate/GED: number analyzed (Participants) | 29 | 32 | 0 | 61
    High school graduate/GED | 12 | 7 |  | 19
    Some college/technical or trade school: number analyzed (Participants) | 29 | 32 | 0 | 61
    Some college/technical or trade school | 7 | 10 |  | 17
    Associate degree: number analyzed (Participants) | 29 | 32 | 0 | 61
    Associate degree | 0 | 4 |  | 4
    Bachelor's degree: number analyzed (Participants) | 29 | 32 | 0 | 61
    Bachelor's degree | 6 | 7 |  | 13
    Professional or graduate degree: number analyzed (Participants) | 29 | 32 | 0 | 61
    Professional or graduate degree | 2 | 1 |  | 3
Employment Status [Count of Participants; unit: Participants] — Population: Employment status data will not be collected from health system participants.
  Participants
    Unemployed/retired: number analyzed (Participants) | 29 | 32 | 0 | 61
    Unemployed/retired | 21 | 16 |  | 37
    Employed Full-time: number analyzed (Participants) | 29 | 32 | 0 | 61
    Employed Full-time | 6 | 9 |  | 15
    Employed Part-time: number analyzed (Participants) | 29 | 32 | 0 | 61
    Employed Part-time | 2 | 6 |  | 8
    Unknown: number analyzed (Participants) | 29 | 32 | 0 | 61
    Unknown | 0 | 1 |  | 1
Subjective Health Status [Count of Participants; unit: Participants] — Population: Subject Health Status data will not be collected from health system participants.
  Participants
    Excellent: number analyzed (Participants) | 29 | 32 | 0 | 61
    Excellent | 1 | 1 |  | 2
    Very good: number analyzed (Participants) | 29 | 32 | 0 | 61
    Very good | 3 | 6 |  | 9
    Good: number analyzed (Participants) | 29 | 32 | 0 | 61
    Good | 14 | 16 |  | 30
    Fair: number analyzed (Participants) | 29 | 32 | 0 | 61
    Fair | 7 | 7 |  | 14
    Poor: number analyzed (Participants) | 29 | 32 | 0 | 61
    Poor | 4 | 2 |  | 6
Subjective Income [Count of Participants; unit: Participants] — Population: Subjective Income data will not be collected from health system participants.
  Participants
    Are comfortable: number analyzed (Participants) | 29 | 32 | 0 | 61
    Are comfortable | 7 | 15 |  | 22
    Have just enough to make ends meet: number analyzed (Participants) | 29 | 32 | 0 | 61
    Have just enough to make ends meet | 14 | 14 |  | 28
    Do NOT have enough to make ends meet: number analyzed (Participants) | 29 | 32 | 0 | 61
    Do NOT have enough to make ends meet | 7 | 3 |  | 10
    Unknown: number analyzed (Participants) | 29 | 32 | 0 | 61
    Unknown | 1 | 0 |  | 1
Difficulty Understanding Written Information [Count of Participants; unit: Participants] — Population: Health literacy data will not be collected from health system participants.
  Participants
    Always: number analyzed (Participants) | 29 | 32 | 0 | 61
    Always | 2 | 0 |  | 2
    Often: number analyzed (Participants) | 29 | 32 | 0 | 61
    Often | 0 | 1 |  | 1
    Sometimes: number analyzed (Participants) | 29 | 32 | 0 | 61
    Sometimes | 7 | 8 |  | 15
    Occasionally: number analyzed (Participants) | 29 | 32 | 0 | 61
    Occasionally | 7 | 5 |  | 12
    Never: number analyzed (Participants) | 29 | 32 | 0 | 61
    Never | 13 | 18 |  | 31
Confidence Filling Out Medical Forms [Count of Participants; unit: Participants] — Population: Health literacy data will not be collected from health system participants.
  Participants
    Extremely: number analyzed (Participants) | 29 | 32 | 0 | 61
    Extremely | 15 | 21 |  | 36
    Quite a bit: number analyzed (Participants) | 29 | 32 | 0 | 61
    Quite a bit | 5 | 5 |  | 10
    Somewhat: number analyzed (Participants) | 29 | 32 | 0 | 61
    Somewhat | 4 | 4 |  | 8
    A little bit: number analyzed (Participants) | 29 | 32 | 0 | 61
    A little bit | 1 | 1 |  | 2
    Not at all: number analyzed (Participants) | 29 | 32 | 0 | 61
    Not at all | 4 | 1 |  | 5
Have Help Reading Hospital Materials [Count of Participants; unit: Participants] — Population: Health literacy data will not be collected from health system participants.
  Participants
    Always: number analyzed (Participants) | 29 | 32 | 0 | 61
    Always | 2 | 0 |  | 2
    Often: number analyzed (Participants) | 29 | 32 | 0 | 61
    Often | 2 | 2 |  | 4
    Sometimes: number analyzed (Participants) | 29 | 32 | 0 | 61
    Sometimes | 4 | 4 |  | 8
    Occasionally: number analyzed (Participants) | 29 | 32 | 0 | 61
    Occasionally | 7 | 6 |  | 13
    Never: number analyzed (Participants) | 29 | 32 | 0 | 61
    Never | 14 | 20 |  | 34
Health System Roles [Count of Participants; unit: Participants] — Population: Health system role data was only collected from health system participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 20 | 20
    Leadership/Administration |  |  | 9 | 9
    Provider (MD, DO, APP) |  |  | 5 | 5
    Clinical Support (MA, RN) |  |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Facilitators and Barriers to Implementing Decision Aids, Provider Notifications, and Personal Risk Calculation Using an Electronic Health Record (EHR) to Promote Colorectal Cancer Screening.
Description: Semi-structured interviews with health system leadership, providers and staff conducted every 3-4 months to discuss facilitators and barriers to implementing decision aids, provider notification, and personal risk calculation using an EHR to promote cancer screening.
Time Frame: 2 years
Population: The initial sample of 8 interviewees identified 12 additional stakeholders, allowing us to "snowball" our sample to complete interviews with 20 participants including primary care providers, nurses, medical assistants, quality and clinic managers, and cancer screening program managers.
Measure: Number; unit: Themes
Arm/Group | Healthcare System Leadership, Providers, and Staff
Number analyzed (Participants) | 20
Themes
  Themes: Barriers identified | 8
  Themes: Facilitators identified | 6

2. Primary Outcome: Challenges and Facilitators of Effective Cancer Screening and Prevention in Primary Care During the COVID-19 Pandemic Among Leadership, Providers, and Staff.
Description: Semi-structured interviews with health system leadership, providers, and staff from the study team's affiliated health systems about their perceptions of the impact of COVID-19 on primary care and cancer screening.
Time Frame: 9 months
Population: 20 leaders, managers, and providers were interviewed in January-July 2021, and 11 were re-interviewed in January-March 2022. We identified five emergent, overarching themes of the impact of COVID-19 pandemic on cancer screening and preventive care services across two healthcare organizations and across the time frame of the COVID-19 pandemic (2020-2022).
Measure: Number; unit: Themes
Arm/Group | Healthcare System Leadership, Providers, and Staff
Number analyzed (Participants) | 20
Themes | 5

3. Primary Outcome: Number of Themes Identified by Patients That Influenced Decisions to Engage in Cancer Screening and Other Healthcare Services, and What Information Was Needed for Making Healthcare Decisions During the COVID-19 Pandemic.
Description: Semi-structured interviews with primary care patients who were due for either breast, cervical, colorectal, or lung cancer screening between April-July 2020 at the study teams affiliate health systems. The interview guide contained questions to explore the patients' understanding, attitudes, and beliefs about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting preventive and other (non-screening) healthcare, and information needed for decision making.
Time Frame: 6 months
Population: We interviewed 32 patients who completed screening in 2020 and 29 patients who did not complete the relevant screening test from April 2020 to the date of the interview.
Measure: Number; unit: Themes
Groups:
- Not Screened Patients: Patients who had at least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020 and did not complete the screening they were selected for at time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
- Screened Patients: Patients who had at least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020 and did complete the screening they were selected for at time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
Arm/Group | Not Screened Patients | Screened Patients
Number analyzed (Participants) | 29 | 32
Themes
  Cancer Screening | 3 | 3
  Other Healthcare Services (non-screening) | 4 | 4
  Health Information | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the interviews. The time frame for patient participants was a one-time phone interview that lasted about 30 minutes. The interviews for health system participants lasted about 30-60 minutes.
Groups:
- Not Screened Patients: Patients who had a least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020 and did NOT complete the screening they were selected for at time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
- Screened Patients: Patients who had a least one primary care visit during the past 24 months at the study team's affiliated health care systems, were due for breast, cervical, colorectal, or lung cancer screening in April-July 2020 and did complete the screening they were selected for at the time of interview.
  Semi-structured interviews-Patients: The interview guide will consist of questions to elicit the patients thoughts about getting preventive healthcare during the COVID-19 pandemic, including perception of risk, barriers to getting healthcare, and information needed for decision making.
Arm/Group | Healthcare System Leadership, Providers, and Staff | Not Screened Patients | Screened Patients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 0/20 | 0/29 | 0/32

LIMITATIONS AND CAVEATS:
We involved just two healthcare systems in one Midwestern city. Our sample of interviewed leaders, providers, and staff may not have been representative of the entire organizations. Our method for identifying patients to interview did not include all patients at these health systems who were due for screening early in the pandemic, so we may have failed to include important perspectives or experiences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT04683744/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT04683744/ICF_001.pdf